CLINICAL TRIAL: NCT01816282
Title: The Use of Fibrin Sealant to Reduce Bleeding After Total Knee Replacement
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Milan (Other)
Responsible Party: Principal Investigator, Pietro Randelli, MD, MD, University of Milan
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Bleeding Control
Record Dates: First submitted 2013-03-15; First posted 2013-03-22 (Estimated); Last update posted 2013-03-25 (Estimated); Status verified 2013-03

CONDITIONS: Total Knee Replacement; Primary Knee Arthroplasty; Osteoarthritis of the Knee
Keywords: TKR; Blood loss; Fibrin Sealant
MeSH Terms: conditions — Osteoarthritis, Knee; Hemorrhage

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Evicel (Experimental)
  Interventions: Drug: Evicel
- Control (No Intervention)

INTERVENTIONS:
Drug: Evicel — Evicel (5ml) is sprayed over the soft tissue after the implant of prosthetic components and before wounding closure
  Arms: Evicel

SUMMARY:
A randomized controlled study is performed to address the question of whether the topical application of a novel fibrin sealant, Evicel (Johnson & Johnson Wound Management, Ethicon, Somerville, NJ) in patient undergoing total knee replacement (TKR) reduce the perioperative blood loss and the need for allogenic blood transfusion compared to a control group. We hypothesize that fibrin sealant decrease the drop in post-operative hemoglobin level after total knee replacement.

DETAILED DESCRIPTION:
Total knee replacement is an invasive surgical procedure that can expose patients to massive perioperative bleeding. This hematic loss results in a high rate of blood transfusion after total knee replacement (TKR) with an incidence from 10% to 58%.Methods to prevent the need for allogenic blood transfusion after TKR include hemodilution, perioperative blood salvage and reinfusion, hypotensive anesthesia, preoperative autologous blood donation and intravenous administration of tranexamic acid.

In the last decade, the topical use of fibrin sealant has become a logical surgical stratagem for reducing blood loss in total knee arthroplasty.Fibrin sealants mimic the final step of the coagulation cascade reducing blood loss and transfusion requirements.

A novel hemostatic agent derived from banked allogenic human plasma (EVICEL, Johnson & Johnson Wound Management, Ethicon, Somerville, NJ) is recently available on the market for a variety of surgical specialty.

A randomized controlled study is conducted to test if the post-operative reduction in hemoglobin level would be lower in the fibrin sealant group compared to a control group.

ELIGIBILITY:
Inclusion Criteria:

* patient scheduled for TKR
* written informed consent
* diagnosis of osteoarthritis

Exclusion Criteria:

* previous intervention on the same Knee (except for meniscectomy)
* Hb pre-operative level lower than 12g/dl for man and 11g/dl for woman
* Anticoagulation therapy or any anti-aggregate treatment not suspended at least 4 days before surgery

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2011-03; Primary Completion 2012-04 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Fall in post-operative hemoglobin level after total knee replacement | First 7 days after surgery
  Hemoglobin values are collected in patients in first week post surgery to assess how these values have changed.

SECONDARY OUTCOMES:
total blood loss | until 7 day after surgery
  Calculation of perioperative blood loss is based on changes in hemoglobin (Hb) level. Assuming that the blood volume V0 on the seventh day after surgery is the same as that before surgery the loss of Hb is estimated according to the following formula:
  Hb-loss (g) =V0 (l)×(Hbpre-op (g/l)-Hb7day post-op(g/l))+Hb-transfused (g) where:
  * Hb-loss (g) is the amount of hemoglobin lost
  * Hbpre-op (g/l) is the hemoglobin level before surgery
  * Hb7day post-op (g/l) is the hemoglobin level in postoperative day 7
  * Hb-transfused (g) is the total amount of allogeneic hemoglobin transfused; a unit of banked blood is considered to contain 52 g of hemoglobin.
  * V0 (l) is the total blood volume of patient and it is calculated using the formula of Nadler:
  V0male(l)=0.3669×height(m)3+0.03219×weight(Kg)+0.6041 V0female(l)=0.3561×height(m)3+0.0338×weight(Kg)+0.1833
  The total blood loss is calculated as follows:
  Blood loss(l)=Hb-loss(g)/Hbpre-op(g/l)
Blood Transfusion rate | until 1 week after Surgery
  Number of patients requiring 1 or more unit of allogenic banked blood

CONTACTS AND LOCATIONS:
Locations (1):
- Unità Operativa Ortopedia e Traumatologia II Policlinico San Donato, San Donato Milanese, Milano, Italy

REFERENCES:
- [Background] Sehat KR, Evans RL, Newman JH. Hidden blood loss following hip and knee arthroplasty. Correct management of blood loss should take hidden loss into account. J Bone Joint Surg Br. 2004 May;86(4):561-5. PMID 15174554
- [Background] Nadler SB, Hidalgo JH, Bloch T. Prediction of blood volume in normal human adults. Surgery. 1962 Feb;51(2):224-32. No abstract available. PMID 21936146
- [Derived] Randelli F, D'Anchise R, Ragone V, Serrao L, Cabitza P, Randelli P. Is the newest fibrin sealant an effective strategy to reduce blood loss after total knee arthroplasty? A randomized controlled study. J Arthroplasty. 2014 Aug;29(8):1516-20. doi: 10.1016/j.arth.2014.02.024. Epub 2014 Feb 26. PMID 24674732